CLINICAL TRIAL: NCT06607198
Title: Clinical-pathological Assessment of Pit-NETs: Data From a Large Multicenter Patients Cohort
Brief Title: Clinical-pathological Evaluation of Pit-NETs
Acronym: PitNET2024
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6859
Record Dates: First submitted 2024-09-17; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Pituitary; Cancer; Neuroendocrine Tumors
MeSH Terms: conditions — Pituitary Diseases; Neoplasms; Neuroendocrine Tumors | interventions — Radiomics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: grading & staging — To investigate the following pathological features of PitNET cell lineage-specific transcription factors, cell type specification by hormone production, proliferative index, p53, mitotic count, expression of somatostatin receptors
Diagnostic Test: PitNET morphology analysis — Revision of the pre-surgical magnetic resonance images (MRIs): tumor maximum diameter, volume, sites of tumor extensions and invasion, and grading of cavernous sinus invasion
Diagnostic Test: Radiomics — To investigate radiomics features of PitNETs
Diagnostic Test: Molecular test: proteomics — To investigate on PitNets of molecular biomarkers Vascular Endothelial Growth Factor (VEGF), Epithelial Growth Factor Receptor (EGFR), somatostatin receptors 1-5 (SSTRs), Fibroblast Growth Factor (FGF), mTOR (mammalian target of rapamycin), Programmed cells Death 1 (PD1) and its ligands (PD-L1), and Cytotoxic T Lymphocyte Associated protein 4 (CTLA4)]

SUMMARY:
Pituitary adenomas, namely pituitary neuroendocrine tumors (PitNETs), are recognized as rare neoplasia by national and international institutions.

Albeit most PitNETs are slow-growing with an indolent behavior, about one-third do not achieve biochemical control, recur, re-grow, and resist conventional treatments.

The predictors of aggressive behavior have not been identified for PitNETs. In 2013 Trouillas and coworkers developed a five tiered clinicopathological score by mixing histopathological data and clinico-radiological evidence of invasion. This system proved of prognostic value. Nonetheless, unlike for NET of gut and lung, no formal grading and/or staging tools were developed. In addition, PitNETs have not been thoroughly investigated by radiomics to predict clinical behavior, nor have druggable pathways been elucidated in PitNET cells to unveil new potential therapeutic approaches.

The first aim of this project is to define grading and staging tools for PitNETs based on: i) lineage-specific transcription factors ; ii) cell type specification by hormone production (prolactin, TSH, LH, FSH, ACTH, GH or none); iii) integration of standard radiological measures with recognized tools for clinical and pathological staging.

The second aim of this project is to investigate radiomics features as predictors of PitNETs behavior, prognosis, and treatment outcome.

The third aim of this project is to investigate whether the expression of molecular biomarkers [Vascular Endothelial Growth Factor (VEGF), Epithelial Growth Factor Receptor (EGFR), somatostatin receptors 1-5 (SSTRs), Fibroblast Growth Factor (FGF), mTOR (mammalian target of rapamycin), Programmed cells Death 1 (PD1) and its ligands (PD-L1), and Cytotoxic T Lymphocyte Associated protein 4 (CTLA4)] may impact on patients prognosis. Identifying new molecular pathways may help fine-tune and schedule the emerging targeted therapies for aggressive PitNETs, including mTOR inhibitors, VEGF, EGFR, and immune check-point inhibitors.

This study will investigate a large multicenter retrospective series of 740 PitNET patients and a prospective cohort of 200 patients to reach these objectives.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients older than 18 years;
* availability of tumor samples for the required pathology analyses;
* clinico-radiological follow-up of at least 5-10 years

Exclusion Criteria:

- Not applicable for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will investigate a large multicenter retrospective series of 740 PitNET patients and a prospective cohort of 200 patients
Sampling Method: Probability Sample
Enrollment: 940 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Grating and staging | 2 years
  To investigate the following pathological features of PitNET cell lineage-specific transcription factors, cell type specification by hormone production, proliferative index, p53, mitotic count, expression of somatostatin receptors, through immunohistochemistry analysis on formalin-fixed paraffin-embedded samples of PitNETs

SECONDARY OUTCOMES:
PitNET morphology analysis | 2 years
  Identification of PitNET morphology features, as tumor maximum diameter, volume, sites of tumor extensions and invasion, and grading of cavernous sinus invasion though the revision of pre-surgical magnetic resonance images
Radiomics | 2 years
  Radiomics features will be extracted and computed using the different standardized methods and platforms for quantitative imaging analysis though different standardized methods and platforms for quantitative imaging analysis. Radiomics analysis will be realized after segmentations test-retest, to evaluate and quantify features' reproducibility.
Molecular test: proteomics | 2 years
  To investigate on PitNets the expression of Vascular Endothelial Growth Factor (VEGF), Epithelial Growth Factor Receptor (EGFR), somatostatin receptors 1-5 (SSTRs), Fibroblast Growth Factor (FGF), mTOR (mammalian target of rapamycin), Programmed cells Death 1 (PD1) and its ligands (PD-L1), and Cytotoxic T Lymphocyte Associated protein 4 (CTLA4)] through proteomic analysis on formalin-fixed paraffin-embedded samples of PitNETs for patients retrospectively included and on frozen tissues for patients prospectively enrolled.

CONTACTS AND LOCATIONS:
Overall Officials: Guido Rindi, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, UOC ANATOMIA PATOLOGICA, Rome, Lazio, Italy